CLINICAL TRIAL: NCT02594956
Title: Impact of the Absence of Nasogastric Decompression After Pancreaticoduodenectomy : A Prospective and Randomized Study
Brief Title: Impact of the Absence of Nasogastric Decompression After Pancreaticoduodenectomy
Acronym: IPOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RennesUH
Record Dates: First submitted 2015-10-29; First posted 2015-11-03 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Digestive System Surgical Procedure; Pancreaticoduodenectomy
Keywords: nasogastric decompression
MeSH Terms: interventions — Enteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- With Nasogastric Decompression (Active Comparator): This group will receive conventional care according to the protocol of the service in place with removal of the nasogastric tube the 3rd postoperative day if the flow is < 500ml / 24h, if not removal will take place on the 5th postoperative day.
  Interventions: Device: nasogastric tube
- Without Nasogastric decompression (Experimental): The nasogastric tube will be take off at the end of the surgery, just after the extubation.
  Interventions: Device: no nasogastric tube

INTERVENTIONS:
Device: no nasogastric tube
  Other Names: no double lumen nasogastric tube
  Arms: Without Nasogastric decompression
Device: nasogastric tube
  Other Names: double lumen nasogastric tube
  Arms: With Nasogastric Decompression

SUMMARY:
The use of nasogastric (NG) decompression after pancreaticoduodenectomy (PD) is a current practice. NG tube is associated with a high rate of morbidity including pulmonary morbidity, delayed gastric emptying and finally an increased length of hospital stay.

The absence of NG decompression could be the corner stone of the concept of the enhanced recovery program after PD.

DETAILED DESCRIPTION:
The use of nasogastric (NG) decompression after pancreaticoduodenectomy (PD) is a current practice. NG tube is associated with a high rate of morbidity including pulmonary morbidity, delayed gastric emptying and finally an increased length of hospital stay. In the era of the enhance recovery after major abdominal surgery, the place of the NG tube remains unproven after PD even if NG tube is clearly abandoned in liver, stomach and colonic surgery. Nowadays, only few retrospective series had reported the feasibility of the absence of nasogastric tube after PD, but not with a randomized control trial. The absence of NG decompression could be the corner stone of the concept of the enhanced recovery program after PD.

The objective of this prospective randomized monocentric study is to evaluate the impact of the absence of NG decompression after PD.

The aim of the study is to decrease postoperative morbidity after PD including pulmonary and delayed gastric emptying complication. The impact of the absence of systematic NG decompression could be interesting in terms of public health with a decreased of length of hospital stay. Furthermore, this is the first randomized study comparing NG tube decompression after PD to absence of NG tube after PD which would bring relevant elements to improve the recovery after PD.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and ≤ 75 years
* patient requiring a PD for benign of malign pathology of the bilio and pancreatic intersection
* patient giving free and informed consent

Exclusion Criteria:

* previous gastric of esophagus surgery
* sever comorbidity such as : end stage renal disease, respiratory failure, heart failure (≥ 3 NYHA)
* Person with a measure of legal protection (guardianship)
* Pregnant woman or nursing mother

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of Clavien and Dindo complication ≥ grade II | up to five days after surgery
  during hospitalisation to demonstrate the feasibility of the absence of NG decompression after pancreaticoduodenectomy

SECONDARY OUTCOMES:
Pulmonary complication | up to 90 days after surgery
  occurrence of pulmonary complication (including atelectasic, pleural effusion, pneumonitis
Gastric emptying | up to five days after surgery
  occurrence of gastric delayed emptying (classified to the ISGPS classification )
Pancreatic fistula | up to 90 days after surgery
  Occurence of pancreatic fistula (classified according to the ISGPS classification)
Food intake | up to five days after surgery
  Time to oral food intake
First gas | up to five days after surgery
  Time to the emission of the first gas
Reinsertion of Nasogastric tube | up to five days after surgery
  NG tube reinsertion rate
Reinsertion of Nasogastric tube | up to five days after surgery
  NG tube reinsertion time
Reinsertion of Nasogastric tube | up to five days after surgery
  NG tube reinsertion for gastroparesis or reintubation
Mortality rate | up to 90 days after surgery
Hospital stay | up to 90 days after surgery
  length of hospital stay
Readmission rate | up to 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Sulpice, MD/PH/prof, Principal Investigator — Rennes UH
Locations (1):
- Centre Hospitalier Universitaire Rennes Pontchaillou, Rennes, France

REFERENCES:
- [Derived] Bergeat D, Merdrignac A, Robin F, Gaignard E, Rayar M, Meunier B, Beloeil H, Boudjema K, Laviolle B, Sulpice L. Nasogastric Decompression vs No Decompression After Pancreaticoduodenectomy: The Randomized Clinical IPOD Trial. JAMA Surg. 2020 Sep 1;155(9):e202291. doi: 10.1001/jamasurg.2020.2291. Epub 2020 Sep 16. PMID 32667635